CLINICAL TRIAL: NCT03298178
Title: ASAN Medical Center Aortic Valve Replacement Registry
Acronym: ASAN-AVR
Status: Active, not recruiting | Type: Observational
Sponsor: Ho-Jin Kim (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Ho-Jin Kim, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV 2017-09
Record Dates: First submitted 2017-09-21; First posted 2017-10-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVR; TAVI; SAVR
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all aortic stenosis
  Interventions: Procedure: TAVR; Procedure: SAVR

INTERVENTIONS:
Procedure: TAVR — All patients who underwent transcatheter aortic valve replacement in Asan medical center, republic of Korea
  Other Names: transcatheter aortic valve replacement
Procedure: SAVR — All patients who underwent surgical aortic valve replacement in Asan medical center, republic of Korea

SUMMARY:
This study evaluates the effectiveness and safety of surgical aortic valve replacement and transcatheter aortic valve replacement in aortic Stenosis.

DETAILED DESCRIPTION:
All TAVR and SAVR cases will be enrolled retrospectively and prospectively.

This registry includes sub group analysis named STRATEGY AS(Role of Sarcopenia and frailTy in pRedicting outcomes After TranscathEter or surGical aortic valve replacement in elderlY patients with Aortic Stenosis: A prospective cohort study). For this sub group analysis, all enrolled subjects will have following tests : EQ-5D, KCCQ-12(Kansas City Cardiomyopathy Questionnaire), ADL(Activities of daily living), IADL(Instrumental. Activities of Daily Living), Nagi & Rosow-Breslau self-reported items, Previous fall events since 6 months (initial) or last visit(F/U), IPAQ(The International Physical Activity Questionnaires), Social frailty screening, CES-D(Center for Epidemiologic Studies Depression Scale), MNA-SF(Mini Nutritional Assessment - Short Form),SPPB score (Short Physical Performance Battery, usual gait speed, balance, chairstand), Multi-task gait test (counting7, animal, motor, motor&counting7), Grip strength, Bioimpedance analysis, Muscle tone at thigh and calf, UEF (Upper extremities function).

ELIGIBILITY:
Inclusion Criteria:

* All successful transcatheter aortic valve replacement or surgical aortic valve replacement
* Written consent

Exclusion Criteria

* Infective endocarditis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All successful transcatheter aortic valve replacement or surgical aortic valve replacement
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
All cause death | 1 year

SECONDARY OUTCOMES:
Cardiovascular mortality | 1,6 and 12 months and 5 years
Cardiovascular mortality | 1,6 and 12 months and 5 years
  Death due to proximate cardiac cause Death caused by noncoronary vascular condition All procedure-related/surgery-related death All valve-related death Sudden or unwitnessed death Death of unknown cause
Myocardial infarction | 1,6 and 12 months and 5 years
Stroke | 1,6 and 12 months and 5 years
  all stroke and TIA
Bleeding | 1,6 and 12 months and 5 years
Operation site complication | 1,6 and 12 months and 5 years
Vascular access site and access-related complication | 1,6 and 12 months and 5 years
Acute kidney injury | at a later date between 30 days or discharge
Event rate of permanent pacemaker insertion | 1,6 and 12 months and 5 years
Other TAVR-related complication | 1,6 and 12 months and 5 years
  Conversion to open surgery Coronary obstruction Mitral valve apparatus damage or dysfunction Cardiac tamponade Endocarditis Valve thrombosis Valve malpositioning TAV-in-TAV deployment(TAV : Transcatheter Aortic Valve)
Prosthetic valve dysfunction | 1,6 and 12 months and 5 years
  Prosthetic aortic valve stenosis Prosthesis-patient mismatch Prosthetic aortic valve regurgitation
Event rate of composite endpoint | 1,6 and 12 months and 5 years
  Device success Early safety within 30 days Clinical efficacy after 30 days defined as death, stroke, valve dysfunction or heart failure requiring hospitalization, severe dyspnea or valve dysfunction NYHA class III or IV
Structural valve deterioration | 1,6 and 12 months and 5 years
Change of NYHA class | 30 days and 1 year
  the New York Heart Association (NYHA) Functional Classification
Change of valve area | 30 days and 1 year
Free from atrial fibrillation | 1,6 and 12 months and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Seung-jung Park, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim HJ, Kang DY, Park H, Ahn JM, Kim JB, Kim SO, Ok YJ, Lee SH, Pyo WK, Ko E, Lee SA, Kim DH, Park SJ, Park DW, Choo SJ. Comparison of Sutureless Bioprosthetic Valve With Surgical or TAVR for Severe Aortic Stenosis. JACC Asia. 2021 Oct 26;1(3):317-329. doi: 10.1016/j.jacasi.2021.08.007. eCollection 2021 Dec. PMID 36341221
- [Derived] Yang Y, Ahn JM, Kang DY, Ko E, Kim S, Kim TO, Kim JH, Lee J, Lee SA, Kim DH, Kim HJ, Kim JB, Choo SJ, Park SJ, Park DW. Implication of Different ECG Left Ventricular Hypertrophy in Patients Undergoing Transcatheter Aortic Valve Replacement. J Am Heart Assoc. 2022 Feb 15;11(4):e023647. doi: 10.1161/JAHA.121.023647. Epub 2022 Feb 3. PMID 35112886
- [Derived] Jeong YJ, Ahn JM, Kang DY, Park H, Ko E, Kim HJ, Kim JB, Choo SJ, Lee SA, Park SJ, Kim DH, Park DW. Incidence, Predictors, and Prognostic Impact of Immediate Improvement in Left Ventricular Systolic Function After Transcatheter Aortic Valve Implantation. Am J Cardiol. 2021 Aug 1;152:99-105. doi: 10.1016/j.amjcard.2021.04.037. Epub 2021 Jun 11. PMID 34127247